CLINICAL TRIAL: NCT00001052
Title: A Phase I, Multicenter, Randomized, Double-Blind, Placebo-Controlled HIV-1 Vaccine Trial to Evaluate the Safety and Immunogenicity of MN Recombinant Soluble gp120/HIV-1 (rsgp120/HIV-1) (Genentech) in Combination With QS21 Adjuvant and/or Alum in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 016A; 10565 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Drug Therapy, Combination; Adjuvants, Immunologic; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections | interventions — Aluminum Hydroxide; saponin QA-21V1

INTERVENTIONS:
Biological: Aluminum hydroxide
Biological: QS-21
Biological: rgp120/HIV-1MN

SUMMARY:
To extend the evaluation of safety and immunogenicity of MN recombinant soluble gp120/HIV-1 (MN rsgp120/HIV-1) in combination with QS21 with or without alum and on two different vaccination schedules.

Recent animal studies indicate that immunizing with MN rsgp120/HIV-1 in combination with QS21 on a 0, 1, 2 month schedule results in a more rapid rise in binding and neutralizing antibody response than on a 0, 1, 6 month schedule. Such an effect may be particularly desirable in vaccine delivery. This study compares these two delivery schedules using the unadjuvanted vaccine formulation rsgp120/HIV-1 with or without addition of alum.

DETAILED DESCRIPTION:
Recent animal studies indicate that immunizing with MN rsgp120/HIV-1 in combination with QS21 on a 0, 1, 2 month schedule results in a more rapid rise in binding and neutralizing antibody response than on a 0, 1, 6 month schedule. Such an effect may be particularly desirable in vaccine delivery. This study compares these two delivery schedules using the unadjuvanted vaccine formulation rsgp120/HIV-1 with or without addition of alum.

Healthy volunteers (20 per group) receive MN rsgp120/HIV-1 (300 or 0 mcg) in combination with QS21 (100 mcg), either with or without alum, at 0, 1, and 2 months or 0, 1, and 6 months. For both vaccination schedules, an additional five volunteers receive only vehicle with alum. The 0 mcg antigen groups are included primarily as negative controls. Subjects may be contacted for follow-up on health status once or twice yearly for at least 5 years.

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* Normal history and physical exam.
* HIV negative by ELISA within 8 weeks of immunization.
* Absolute CD4 count >= 400 cells/mm3.
* Normal urine dipstick with esterase and nitrite.

Exclusion Criteria

Co-existing Condition:

Subjects with the following symptoms or conditions are excluded:

* Hepatitis B surface antigen.
* Medical or psychiatric condition (such as recent suicidal ideation or present psychosis) that precludes compliance.
* Occupational responsibilities that preclude compliance.
* Active syphilis. NOTE: Subjects with serology documented to be false positive or due to a remote (> 6 months) treated infection are eligible.
* Active tuberculosis. NOTE: Subjects with a positive PPD and normal chest x-ray showing no evidence of TB and not requiring isoniazid therapy are eligible.

Subjects with the following prior conditions are excluded:

* History of immunodeficiency, autoimmune disease, or use of immunosuppressive medications.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* History of allergy to thimerosal.
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension).
* Prior psychiatric condition (such as history of suicide attempts or past psychosis) that precludes compliance.
* History of cancer unless there has been surgical excision that is considered to have achieved cure.

Prior Medication:

Excluded:

* Live attenuated vaccines within 60 days prior to study entry. (NOTE: Medically indicated subunit or killed vaccines, such as influenza or pneumococcal, are allowed but should be given at least 2 weeks prior to HIV immunizations.)
* Experimental agents within 30 days prior to study entry.
* Prior HIV vaccines.

Prior Treatment:

Excluded:

* Receipt of blood products or immunoglobulin within the past 6 months.

Risk Behavior:

* Subjects are NOT excluded on the basis of HIV risk behaviors, but AVOIDANCE of any activity that may expose subject to HIV (e.g., unprotected sex or needle sharing) is STRONGLY RECOMMENDED.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Study Completion 1997-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: McElrath J, Study Chair
Locations (5):
- United States (5):
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York
  - JHU AVEG, Pittsburgh, Pennsylvania
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Zolla-Pazner S, Alving C, Belshe R, Berman P, Burda S, Chigurupati P, Clements ML, Duliege AM, Excler JL, Hioe C, Kahn J, McElrath MJ, Sharpe S, Sinangil F, Steimer K, Walker MC, Wassef N, Xu S. Neutralization of a clade B primary isolate by sera from human immunodeficiency virus-uninfected recipients of candidate AIDS vaccines. J Infect Dis. 1997 Apr;175(4):764-74. doi: 10.1086/513969. PMID 9086128
- [Background] Evans TG, McElrath MJ, Matthews T, Montefiori D, Weinhold K, Wolff M, Keefer MC, Kallas EG, Corey L, Gorse GJ, Belshe R, Graham BS, Spearman PW, Schwartz D, Mulligan MJ, Goepfert P, Fast P, Berman P, Powell M, Francis D; NIAID AIDS Vaccine Evaluation Group. QS-21 promotes an adjuvant effect allowing for reduced antigen dose during HIV-1 envelope subunit immunization in humans. Vaccine. 2001 Feb 28;19(15-16):2080-91. doi: 10.1016/s0264-410x(00)00415-1. PMID 11228380